CLINICAL TRIAL: NCT07013240
Title: Immediate Post-surgical Botulinum Toxin Injections to Prevent Dystrophic Scars After Sternotomy : a Placebo-controlled Randomized Clinical Trial
Brief Title: Botulinum Toxin Injection After Sternotomies to Improve Scar Aspect and Impact
Acronym: BotuCiSter
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHUBX 2024/31
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Sternotomy Closure,Open Heart Surgery
Keywords: scar; keloid; botulinum toxin; sternotomy
MeSH Terms: conditions — Cicatrix; Keloid | interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the Methodology Center and the Bordeaux University Hospital Pharmacy will have access to the correspondence list between the patient's number, the type of product and the area treated (lower or upper part of the scar). At no time during the study will investigators or patients have access to this list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upper Arm (Experimental): Intervention (botulinum toxin) in the upper half of the scar and placebo in the lower half
  Interventions: Drug: Botulinum toxin injection
- Lower Arm (Experimental): Intervention (botulinum toxin) in the lower half of the scar, and placebo in the upper half.
  Interventions: Drug: Botulinum toxin injection

INTERVENTIONS:
Drug: Botulinum toxin injection — Intervention will be made immediately after surgery, still under general anesthesia, by the cardiac surgeon, after suture.
  Each patient will receive (either in the lower part or the upper part of the scar according to randomization) 50 international units (IU) of type A botulinum toxin (Botox®, Allergan aesthetics) diluted in 1 mL of saline to enable injection of 5 IU at each point, every centimeter, at 1 cm of each scar side.
  An equivalent volume of saline will be injected under the same modalities in the other part of the scar.

SUMMARY:
Sternotomy scars, which are localized in a high-tension area are often dystrophic, hypertrophic or keloidal, and can be difficult to accept to patients who already endured a heavy intervention with high psychologic impact. The investigators wish to evaluate immediate post-surgical injection of botulinum toxin to improve scar aspect and impact. A randomized, placebo-controlled, split-scar clinical trial will determine the improvement of scar aspects assessed by standardized scores (SBSES, POSAS), patient satisfaction and tolerance.

DETAILED DESCRIPTION:
Adult wound healing does not restore the original skin architecture, and results in fibrotic scars. Specifically in high-tension areas and due to activation of fibrogenesis pathways, wound healing processes can lead to pathological scarring, hypertrophic scars, or keloids. The anterior thoracic region is one the body area suggested to the highest tensions, and sternotomies are performed perpendicularly to the lines of skin tension. Therefore, sternotomy scars are often dystrophic, inaesthetic and fibrous, or even hypertrophic. Depending on geographical distribution, sternotomy scars are found hypertrophic in 10 % to more than 50 % of cases. Aesthetic impact or related symptoms such as pruritus and pain impair psychological state and alter quality of life of these patients who endured a frequently difficult to handle surgical procedure.

Botulinum toxin type A is a neurotoxin derived from Clostridium botulinum culture. Through inhibition of pre-synaptic acetylcholine release, it induces local muscle paralysis that is reversible in a few months. Its interest is widely described in urology and neurology. Its dermatologic uses include the cosmetic purpose to reduce face wrinkles and the functional purpose to reduce hyperhidrosis. Its safety is well established. It has been proposed in the prevention and treatment of hypertrophic scars and keloids, and has been shown to reduce TGFß1, a main actor of fibrogenesis and pathological scarring. Through reduction of myofibroblastic differentiation, it downregulates mechanisms leading to dystrophic scars.

It was proposed in the improve scar aspect after surgical procedures, and early post-operative local injections showed efficacy in thyroidectomies, mammoplasties, or face surgeries to enhance scar aspect. Regarding sternotomy, a single study in China with a small sample (17 patients) studied post-operative injections (8 to 14 days after) of botulinum toxin. This split-scar study reported significant improvement of Vancouver Scar Scale, scar width and patient satisfaction in the treated site, at 6 months.

The authors aim to evaluate immediate post-operative botulinum toxin after sternotomies, to improve scar aspect through standardized scores (Stony Brook Scar Evaluation Scale, Patient and Observer Scar Assessment Scale) and impact through patient satisfaction at 6 and 18 months. The double-blind randomized placebo-controlled trial will be conducted in split-scar method, with administration for each patient of treatment (botulinum toxin) or placebo (saline) in the upper or lower part of scar, according to randomization.

Each patient will serve as its own control and will be evaluated for up to 18 months by a dermatological team, following standardized monitoring, including objective and subjective scores, as well as tolerance data.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Scheduled sternotomy at Bordeaux University Hospital within the next 4 months
* Person affiliated with or benefiting from a social security system
* Patient able to attend follow-up visits required by the study
* Free, informed, and written consent signed by the participant or an impartial witness (in case the participant is unable to write) and the investigator (no later than the day of inclusion)

Exclusion Criteria:

* Known allergy to botulinum toxin type A or any excipient in BOTOX® (human albumin, sodium chloride)
* Neuromuscular transmission disorder (myasthenia gravis or Lambert-Eaton syndrome)
* Motor peripheral neuropathy (such as amyotrophic lateral sclerosis or motor neuropathy)
* Infection at the injection sites
* Pregnancy or breastfeeding
* Person under protection measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-05 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Stony Brooke Scar Scale score | Month 6
  The Stony Brook Scar Evaluation Scale (SBSES) was developed by Singer et al. in 2007. It is based on five scar indicators: width, elevation or depression, color, suture or staple marks, and overall appearance.Each indicator is assigned a score between 0 and 5 points. These scores are totaled to obtain the final score between 0 and 5 points. This score will be determined for each half of scar (superior part and inferior part).

SECONDARY OUTCOMES:
Measure of scar width in millimeters | Month 3, month 6, month 12 and month 18
Evaluation of scar with POSAS : observer scale | Month 3, month 6, month 12 and month 18
  The observer's POSAS scale comprises six parameters (vascularity, pigmentation, thickness, relief, elasticity and surface).
  Each parameter is rated on a scale from 1 ("normal skin") to 10 ("worst scar imaginable").
  The sum of the six parameters constitutes the observer's total POSAS score scale .
  In addition, a general opinion is scored from 1 to 10. All parameters should preferably be compared to normal skin on a comparable a comparable anatomical region.
  This scale will be determined for each half of scar (superior part and inferior part).
Evaluation of scar with The Physician's Global Assesment (PGA) | Month 3, Month 6, Month 12 and Month 18
  The Physician's Global Assesment (PGA) evaluates the scar based on whether it is considered an Invisible scar ; a Scar as fine as a pencil line, of a color similar to the adjacent skin ; a Visible scar, little infiltrated or flat, discreetly colored ; a Widened and infiltrated scar, visible suture lines, of a color contrasting with the skin ; a Hypertrophic scar, raised, hypervascularized or very hyperpigmented ; a Keloid.
  This evaluation will be determined for each half of scar (superior part and inferior part).
Evaluation of Stony Brooke Scar Scale score | Month 3, Month 12 and Month 18
  The Stony Brook Scar Evaluation Scale (SBSES) was developed by Singer et al. in 2007. It is based on five scar indicators: width, elevation or depression, color, suture or staple marks, and overall appearance. Each indicator is assigned a score between 0 and 1 point. These scores are totaled to obtain the final score between 0 and 5 points.
  This scale will be determined for each half of scar (superior part and inferior part).
Evaluation of scar with POSAS : Patient scale | Month 3, Month 6, Month 12 and Month 18
  The patient's POSAS scale comprises six parameters (pain, itching, color, stiffness, thickness and irregularity).
  Each parameter is rated on a scale from 1 ("normal skin") to 10 ("worst scar imaginable").
  In addition, a general opinion is scored from 1 to 10. The sum of all these parameters constitutes the patient's total POSAS score scale.
  All parameters should preferably be compared to normal skin on a comparable a comparable anatomical region.
  This evaluation will be determined for each half of scar (superior part and inferior part).
Satisfaction numerical scale | Month 3, Month 6, Month 12 and Month 18
  Scar satisfaction is rated on a scale from 0 ("not at all satisfied") to 10 ("extremely satisfied").
  This scale will be determined for each half of scar (superior part and inferior part).

CONTACTS AND LOCATIONS:
Overall Officials: Robin ZAGALA, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Yes
The data is available from Dr ZAGALA. An email can be sent to her so that she can contact the data manager and owner, the Bordeaux University Hospital. The data can be made available after contractual agreement.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Singer AJ, Arora B, Dagum A, Valentine S, Hollander JE. Development and validation of a novel scar evaluation scale. Plast Reconstr Surg. 2007 Dec;120(7):1892-1897. doi: 10.1097/01.prs.0000287275.15511.10. PMID 18090752